CLINICAL TRIAL: NCT05660213
Title: A Multicenter Registry Study on the Efficacy and Safety of Different Treatment Regimens for Unresectable CNLC Liver Cancer Stage III Hepatocellular Carcinoma
Brief Title: A Multicenter Registry Study on Stage III Hepatocellular Carcinoma in Unresectable CNLC Liver Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jia Fan, Professor, Fudan University
Other Study IDs: HELICOP
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Huaier granules; Unresectable hepatocellular carcinoma; curative effect; safety; Anti-PD-1/PD-L1 antibody drugs
MeSH Terms: interventions — Immunotherapy; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort A: Targeted drugs combined with anti-PD-1 / PD-L1 antibodies
  Interventions: Drug: Targeted drugs combined with anti-PD-1/PD-L1 antibodies
- Cohort B: TACE (transarterial chemoembolization) combined with target immunotherapy
  Interventions: Drug: TACE (transarterial chemoembolization) combined with targeted/immunotherapy
- Cohort C: Lenvatinib monotherapy
  Interventions: Drug: Lenvatinib monotherapy
- Cohort D: Huaier granules combined with any of the above Cohorts for treatment
  Interventions: Drug: Huaier granules combined with any of the above Cohorts for treatment

INTERVENTIONS:
Drug: Targeted drugs combined with anti-PD-1/PD-L1 antibodies — Targeted drugs combined with anti-PD-1/PD-L1 antibodies
  Groups: Cohort A
Drug: TACE (transarterial chemoembolization) combined with targeted/immunotherapy — TACE (transarterial chemoembolization) combined with targeted/immunotherapy
  Groups: Cohort B
Drug: Lenvatinib monotherapy — For patients weighing less than 60 kg, the recommended daily dose of this product is 8 mg (2 capsules of 4 mg), once daily; For patients weighing ≥ 60 kg, the recommended daily dose of this product is 12 mg (3 capsules of 4 mg), once daily. Treatment should be continued until disease progression or intolerable toxic reactions occur.
  Groups: Cohort C
Drug: Huaier granules combined with any of the above Cohorts for treatment — Oral administration of Huaier granules, 10g each time, 3 times a day, until the end of the study, intolerable toxicity, withdrawal from the study for any reason, or death, whichever occurs first; Or the researcher determines that there is no longer any benefit.It is recommended that the date of first use of Huaier granules be determined by the researchers, and after disease progression, the researchers and patients should jointly decide whether to continue receiving Huaier granules treatment.
  Other Names: Z20000109#NMPA Approval Number#
  Groups: Cohort D

SUMMARY:
This study is a multicenter, registered research aimed at evaluating the efficacy of different treatment regimens in the treatment of unresectable CNLC liver cancer stage III hepatocellular carcinoma

DETAILED DESCRIPTION:
This study is a multicenter, observational, natural cohort registration study. We plan to continuously include 750 subjects diagnosed with unresectable CNLC stage III hepatocellular carcinoma (HCC) at selected research centers. According to the actual clinical diagnosis and treatment plan of patients, the following treatment modes will be included in the Cohort of patients:

Cohort A: Targeted drugs combined with anti-PD-1/PD-L1 antibodies Cohort B: TACE (transarterial chemoembolization) combined with targeted/immunotherapy Cohort C: Lenvatinib monotherapy Cohort D: Huaier granules combined with any of the above Cohorts for treatment Throughout the entire study period, it is planned to recruit patients who have visited the selected research center within 12 months (December 2024 to December 2025). Each individual subject will be followed up every 8 weeks until the diagnosis and treatment mode changes, disease progression progresses, or the patient withdraws from the study or dies for any reason, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

·≥ 18 years old;

* Diagnosed as unresectable hepatocellular carcinoma through histopathological and/or cytological examination, or meeting the clinical diagnostic criteria for hepatocellular carcinoma in the 2022 edition of the guidelines for the diagnosis and treatment of primary liver cancer;
* CNLC liver cancer stage III;
* Liver function Child Pugh A or B grade 7 points;
* Has not received systematic treatment in the past;
* Patients with active HBV infection who meet one of the following conditions can be enrolled: ① Within 28 days before enrollment, the patient's HBV DNA is less than 500 IU/mL. If they have received anti HBV treatment, they need to continue their original antiviral treatment; If anti HBV treatment has not been received, it is necessary to receive anti HBV treatment throughout the entire course of medication (according to local treatment standards; for example, entecavir); ② For patients with HBV DNA>500 IU/mL and who have not received antiviral therapy, they must receive at least 7 days of antiviral therapy (according to local treatment standards; for example, entecavir) before enrollment in this study, and are willing to continue receiving antiviral therapy during the study. Before enrollment, the serum HBV-DNA virus should be retested to decrease by more than 1 log value For patients with HBV DNA>500 IU/mL and who have received antiviral therapy, they must receive at least 7 days of antiviral therapy (according to local treatment standards; for example, entecavir) before enrollment in this study, and are willing to continue receiving antiviral therapy during the study. Serum HBV-DNA virus levels should be retested before enrollment;
* Active HCV infected individuals with stable disease status after treatment;
* At least one tumor lesion available for evaluation;
* Clear consciousness, language expression ability or reading ability, able to communicate normally, and cooperate to complete the questionnaire evaluation;
* Voluntarily join this study and sign an informed consent form.

Exclusion Criteria:

* Simultaneously having two or more active primary malignant tumors;
* Portal vein cancer thrombus invades the superior mesenteric vein;
* Received radiation therapy within the past 4 weeks;
* Expected survival time is less than 3 months;
* Pregnant or lactating women or those planning to conceive;
* Coagulation dysfunction (INR>2.0, PT>16 s) or diseases with a strong likelihood of bleeding (including but not limited to esophageal and/or gastric variceal bleeding, active ulcers, uncontrolled hypertension);
* Refusing to cooperate with follow-up visits;
* Other reasons led the researchers to believe that it was not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the whole study period, a total of 750 patients in the selected research centers from December 2024 to December 2025 were planned to be recruited consecutively, including 150 in cohort a, 150 in cohort B, 150 in cohort C, and 300 in cohort D. A single subject was visited every 8 weeks after enrollment until the diagnosis and treatment mode changed, disease progression or the patient withdrew from the study or died for any reason, whichever occurred first. The maximum duration of a single subject's total visit shall not exceed 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
ORRObjective response rate (ORR) | start of treatment until 24-month follow-up
  It defined as the proportion of subjects who achieve complete response (CR) or partial response (PR) in primary tumor imaging evaluation.
Progression free survival (PFS) | Start of treatment until 24-month follow-up
  It defined as the time from the date the subject first receives combination therapy until the first observation of tumor progression or death from any cause.
Disease control rate (DCR) | Start of treatment until 24-month follow-up
  It defined as the proportion of subjects who achieve complete response (CR), partial response (PR), or disease stability (SD) as assessed by primary tumor imaging.
Time to Response（TTR） | Start of treatment until 24-month follow-up
  It defined as the time from the date the subject first receives combination therapy to the first observation of tumor response (CR or PR).
Duration of Response (DoR) | Start of treatment until 24-month follow-up
  It defined as the time from the first observation of tumor remission (CR or PR) in a subject receiving combination therapy to the first observation of tumor progression or death from any cause.
Overall survival (OS): | Start of treatment until 24-month follow-up
  It defined as the time from the day of randomization of patients to death from any cause.

SECONDARY OUTCOMES:
Quality of Life Score | Start of treatment until 24-month follow-up
  Evaluation using the EORTC QLQ-C30 (Chinese version) core quality of life scale developed by the European Organization for Cancer Research and Treatment.
The incidence and severity of adverse events (AE) and severe adverse events (SAE) | Start of treatment until 24-month follow-up
  The definition and severity grading of AE and SAE refer to the corresponding descriptions in the definition and evaluation section of adverse events, and the incidence rate is defined as the proportion of patients with AE and SAE to the corresponding total population.
The incidence and severity of adverse reactions (ADR), severe adverse reactions (SADR), suspicious and unexpected severe adverse reactions (SUSAR) | Start of treatment until 24-month follow-up
  The definition and severity grading of ADR, severe ADR, and SUSAR refer to the corresponding descriptions in the definition and evaluation section of adverse events. The incidence rate is defined as the proportion of patients with ADR, severe ADR, and SUSAR to the corresponding total population.
The incidence and severity of Adverse Events of Special Concern (AESI) | Start of treatment until 24-month follow-up
  AESI includes proteinuria, enteritis, and immune-mediated myocarditis. The incidence is defined as the proportion of patients who experience AESI to the corresponding total population, and the severity grading refers to the corresponding description in the definition and evaluation section of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, PhD, Principal Investigator — Affiliated Zhongshan Hospital, Fudan University

IPD SHARING:
Plan to Share IPD: No